CLINICAL TRIAL: NCT05358457
Title: Pilot Study to Evaluate the Effectiveness of Online Familiar Metacognitive Training (MCTf) in Mothers With Psychosis and Their Adolescent Children
Brief Title: Pilot Study to Evaluate the Effectiveness of Online Familiar Metacognitive Training (MCTf)
Acronym: MCTf
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Fundació Sant Joan de Déu (Other)
Collaborators: Parc Sanitari Sant Joan de Déu (Other); Hospital de Sant Pau (Other); Institut Pere Mata (Unknown); Parc Taulí Hospital Universitari (Other); Hospital de Mataró (Other); Centre d'Higiene Mental Les Corts (Other); Instituto de Investigación Sanitaria de la Fundación Jiménez Díaz (Other); Hospital del Mar (Other); Hospital Universitario Marqués de Valdecilla (Other); Hospitales Universitarios Virgen del Rocío (Other); Fundació Vidal i Barraquer (Unknown); Hospital Sant Joan de Deu (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PI21/00012
Record Dates: First submitted 2022-04-01; First posted 2022-05-03 (Actual); Last update posted 2022-05-03 (Actual); Status verified 2022-04

CONDITIONS: Psychosis; Mother-Child Relations
MeSH Terms: conditions — Psychotic Disorders

STUDY DESIGN:
Intervention Model Description: Parrallel Assigment. This is a randomized clinical trial in which some patients receive the MCTf intervention and others treatment as usual
Who Masked: Outcomes Assessor
Masking Description: The evaluator will be blind to the group that ows the patients included
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Online Familiar Metacognitive Training (Experimental): Metacognitive training for psychosis. The MCTf consists of 11 therapeutic units developed during weekly sessions lasting 45 and 60 minutes. Each unit contains abundant therapeutic material that includes psychoeducational information, exercises and case examples.The group will be composed of 3-4 mothers with psychosis and her adolescent children and two therapists. The application of the intervention will be by a secure videoconfering method.
  Interventions: Behavioral: Familiar Metacognitive Training
- Control group (No Intervention): The control group will be receive treatment as usual (TAU).

INTERVENTIONS:
Behavioral: Familiar Metacognitive Training — The original metacognitive training program consist of 8 therapeutic units and 2 complementary. Seven of the therapeutic units address cognitive deviations and errors that are frequently seen in problem solving in schizophrenia, involved in the formation and maintenance of delusions. The other three units work with metacognition and the aims of the progra, as a psychoeducation session, so in total the MCTf will include 11 sessions.
  Arms: Online Familiar Metacognitive Training

SUMMARY:
The objective of this study is to adapt and evaluate the efficacy of Familiar Metacognitive Training (MCTf) in mothers and adolescent children in a group context with the main purpose of improving family relationships, cognitive awareness and symptoms of women with psychosis and the knowledge of the disease by the children. Secondary objectives: to evaluate the improvement in metacognition and social cognition, symptoms, protective factors and self-perception of stigma.

DETAILED DESCRIPTION:
This is a randomized clinical trial will be carried out in which a group of mothers with psychosis and their adolescent children (between 12 and 18 years old) will receive the MCTf online and the other group will receive the treatment as usual. In total, 48 mothers and their children will be recruited from a total of 11 adult mental health care centers. Mothers will be evaluated with cognitive insight scales, other metacognitive and social cognition scales, symptoms, family and social functioning, protective factors (self-steem, resilience, and coping strategies) and self-perceived stigma. The adolescent children will be evaluated with symptoms, metacognition and social cognition, family and social functioning, knowledge of the mother´s illness and protective factors scales. The will be assessed at 2 times: baseline and post-therapy. The Metacognitive training is a group psychological intervention that has demonstrated its efficacy in improve symptoms, insight, metacognition and cognition in people with psychosis. Our hypothesis is that MCTf will be help the adolescents to better understand their mother´s thoughts and their understanding of metacognition and, consequently, to decrease anxiety and depressive symptoms.Furthermore, the investigators expect an increase in familiar and social functioning, as well as in protective factors such as: self-steem, resilience and coping strategies.

ELIGIBILITY:
Inclusion Criteria:

* Presence of one of the following diagnoses according to DSM-V criteria: schizophrenia, unspecific psychotic disorder, schizoaffective disorder, delusional disorder, brief psychotic disorder, schizophreniform disorder.
* Mother of one o more adolescent (12-18 years old).
* Psychopatological stability in the previous 3 months.(without medication changes).

Exclusion Criteria:

* Head injury or intellectual disabillity (premorbid IQ <=70)
* Present scores on the PANSS >= hostility, lack of cooperation or suspiciousness, to guarantee a good relationship in the group.
* Patients with substance dependence disorder.

Inclusion/exclusion criteria of adolescents are: 1.age between 12 and 18 yerars old, 2. interested in the group. Exclusion criteria: Head injury or intellectual disabillity (premorbid IQ <=70).

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes
Enrollment: 48 (Estimated)
Dates: Start 2022-09 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
BCIS Beck Cognitive and Insight Scale (Beck et al., 2004; Gutierrez-Zotes et al., 2012) | baseline
  This scales is a self-registering measure of 15 items. It has 2 dimensions:self-reflection and self-certaintly. A compound index of cognitive insight is obtained as the substraction of self-certaintly from self-reflection.Range 0-45. Higher values represent a better outcome.
BCIS Beck Cognitive and Insight Scale (Beck et al., 2004; Gutierrez-Zotes et al., 2012) | up to 11 weeks
  This scales is a self-registering measure of 15 items. It has 2 dimensions:self-reflection and self-certaintly. A compound index of cognitive insight is obtained as the substraction of self-certaintly from self-reflection.Range 0-45. Higher values represent a better outcome.

SECONDARY OUTCOMES:
CBQ Cognitive Biais Questionnaire (Peters et al., 2013; Guiterrez-Zotes et al.,2021 | baseline
  Scale for the assessment of the most cognitive biases in psychosis.Higher values represent more biases.
CBQ Cognitive Biais Questionnaire (Peters et al., 2013; Guiterrez-Zotes et al.,2021 | up to 11 weeks
  Scale for the assessment of the most cognitive biases in psychosis. Higher values represent more biases.
Jumping to conclusions (Garety et al., 1991; Dudley et al., 1997) | baseline
  Scale for the assessment to the Jumping to conclusions bias. 3 tasks will be included. JTC is considered if the decision is taken before the third ball.
Jumping to conclusions (Garety et al., 1991; Dudley et al., 1997) | up to 11 weeks
  Scale for the assessment to the Jumping to conclusions bias. 3 tasks will be included. JTC is considered if the decision is taken before the third ball.
IPSAQ, Internal, personal and situational Attributions Questionnaire.(Bentall et al., 1991; Diez-Alegria, 2006) | baseline
  The scale assess the attributional style in different situations.There are no ranges.
IPSAQ, Internal, personal and situational Attributions Questionnaire.(Bentall et al., 1991; Diez-Alegria, 2006) | up to 11 weeks
  The scale assess the attributional style in different situations.There are no ranges.
The Hinting Task (Corcoran et al., 1995; Gil et al., 2012) | baseline
  The scale asses Theory of Mind. Possible Range 0-12. Higher values represent a better outcome.
The Hinting Task (Corcoran et al., 1995; Gil et al., 2012) | up to 11 weeks
  The scale asses Theory of Mind. Possible Range 0-12. Higher values represent a better outcome.
Face Test (Baron Cohen, 1997; Huerta-Ramos et al., 2021) | baseline
  20 photographs that express ten basic and ten complex emotions. Possible range 0-20. Higher values representa better outcome.
Face Test (Baron Cohen, 1997; Huerta-Ramos et al., 2021) | after the intervention
  20 photographs that express ten basic and ten complex emotions. Possible range 0-20. Higher values representa better outcome.
SFRT-2 .Situational feature recognition test 2 (Gomez-Gastiasoro et al., 2018) | baseline
  The scales assess social perception. There are no ranges
SFRT-2 .Situational feature recognition test 2 (Gomez-Gastiasoro et al., 2018) | up to 11 weeks
  The scales assess social perception. There are no ranges
FES Family Enviromental Scale (Moos et al., 1987; Fernandez-Ballesteros., 1995) | baseline
  The scale include 3 dimensions: relationships, development and stability.
FES Family Enviromental Scale (Moos et al., 1987; Fernandez-Ballesteros., 1995) | up to 11 weeks
  The scale include 3 dimensions: relationships, development and stability.
SWLS Satisfaction with life style (Pons et al., 2002) | baseline
  The scale asses the degree of satisfaction of the person with their life in 5 items. Self-administered.
SWLS Satisfaction with life style (Pons et al., 2002) | up to 11 weeks
  The scale asses the degree of satisfaction of the person with their life in 5 items. Self-administered.
PANSS.Positive and Negative Syndrome Scale (Kay et al., 1987; Peralta and Cuesta., 1994) | baseline
  This scale measure 30 symptoms on a scale 1-7, with higher scores indicating greater psychopathology
PANSS.Positive and Negative Syndrome Scale (Kay et al., 1987; Peralta and Cuesta., 1994) | up to 11 weeks
  This scale measure 30 symptoms on a scale 1-7, with higher scores indicating greater psychopathology
CDSS. Calgary Depression Scale for Schizophrenia (Addington et al., 1990) | baseline
  The scale assess affective symptoms. Higher values indicate more symptoms.
CDSS. Calgary Depression Scale for Schizophrenia (Addington et al., 1990) | up to 11 weeks
  The scale assess affective symptoms. Higher values indicate more symptoms.
SUMD. Scale of Unaweressness of Mental Disorder (Amador., 1993; Ruiz et al., 2008) | baseline
  The scale assess awareness of illness in people with schizophrenia, according to the evaluator´s vision
SUMD. Scale of Unaweressness of Mental Disorder (Amador., 1993; Ruiz et al., 2008) | up to 11 weeks
  The scale assess awareness of illness in people with schizophrenia, according to the evaluator´s vision
EEAG-Scale of Functioning (Endicot et al., 1976) | baseline
  This scale measures the general functioning of the patient on a scale that ranges from 0 to 100.
EEAG-Scale of Functioning (Endicot et al., 1976) | up to 11 weeks
  This scale measures the general functioning of the patient on a scale that ranges from 0 to 100.
Rosenberg Self-Esteem Scale (Martín Albó et al., 2007) | baseline
  Questionnaire to explore personal self-esteem understood as feelings of personal worth and self-respect. The scale consist of 10 items.
Rosenberg Self-Esteem Scale (Martín Albó et al., 2007) | up to 11 weeks
  Questionnaire to explore personal self-esteem understood as feelings of personal worth and self-respect. The scale consist of 10 items.
CD Risk 17 (Serrano et al., 2013) | baseline
  The scale assess resilience with a total of 17 items.
Coping Strategies Inventory (Tolbin et al., 1989; Cano et al; 2007) | baseline
  The scale includes 8 scales that assess the frequency of use of primary coping strategies and the perception of coping self-efficacy.
Coping Strategies Inventory (Tolbin et al., 1989; Cano et al; 2007) | up to 11 weeks
  The scale includes 8 scales that assess the frequency of use of primary coping strategies and the perception of coping self-efficacy.
SSQ Self Stigma Questionnaire (Ochoa et al.,2015) | baseline
  The scales assess self-stigma. It consists of 14 items and is self-administered
SSQ Self Stigma Questionnaire (Ochoa et al.,2015) | up to 11 weeks
  The scales assess self-stigma. It consists of 14 items and is self-administered
PAM Psychosis Attachment Measure (Berry et al., 2006; Sheinbaum et al., 2013) | baseline
  The scale assess attachment styles
CTQ-SF Childhood Trauma Questionnaire (Bernstein et al., 1994; Hernández et al., 2012) | baseline
  The self-report includes a 28-item test that measures 5 types of maltreatment - emotional, physical, and sexual abuse, and emotional and physical neglect.
YSR Youth Self-Report (Achembach., 1991; Lemos et al., 2002) | baseline
  It is an instrument to assess symptoms in adolescents between 11 and 18 years old.
YSR Youth Self-Report (Achembach., 1991; Lemos et al., 2002) | up to 11 weeks
  It is an instrument to assess symptoms in adolescents between 11 and 18 years old.
KASI The Knowledge About Schizophrenia Interview | baseline
  Scale to asses the beliefs of the disorder
KASI The Knowledge About Schizophrenia Interview | up to 11 weeks
  Scale to asses the beliefs of the disorder

OTHER OUTCOMES:
WAIS-IV (Weschler Adults Intelligence Scale, 1955) | baseline
  vocabulary subscale to explore premorbid IQ
TMT-A Trail Making Test, Retain, 1993 | baseline
  Visual attention and task switching. Higher values represent a worse outcome.
TMT-A Trail Making Test, Retain, 1993 | up to 11 weeks
  Visual attention and task switching. Higher values represent a worse outcome.
TMT-B Trail Making Test, Retain, 1993 | baseline
  Visual attention and task switching. Higher values represent a worse outcome.
TMT-B Trail Making Test, Retain, 1993 | up to 11 weeks
  Visual attention and task switching. Higher values represent a worse outcome.
WAIS-IV (Weschler Adults Intelligence Scale, 1955) | baseline
  Digits subscale. Higher values represent a better outcome.
WAIS-IV (Weschler Adults Intelligence Scale, 1955) | up to 11 weeks
  Digits subscale. Higher values represent a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Susana Ochoa, Phd, Principal Investigator — Parc Sanitari Sant Joan de Deu

REFERENCES:
- [Derived] Ochoa S, Espinosa V, Lopez-Carrilero R, Martinez I, Barrera AH, Birules I, Barajas A, Pelaez T, Diaz-Cutraro L, Coromina M, Gonzalez-Rodriguez A, Verdaguer-Rodriguez M, Gutierrez-Zotes A, Palma-Sevillano C, Montes C, Gallego J, Paya B, Casanovas F, Roldan M, Noval E, Varela Casals P, Salas-Sender M, Aznar A, Ayesa-Arriola R, Pousa E, Canal-Rivero M, Garrido-Torres N, Montserrat C, Munoz-Lorenzo L, Crosas JM. Effectiveness of family metacognitive training in mothers with psychosis and their adolescent children: a multicenter study protocol. Front Psychol. 2024 Mar 22;15:1359693. doi: 10.3389/fpsyg.2024.1359693. eCollection 2024. PMID 38586292